CLINICAL TRIAL: NCT07232212
Title: Survival Outcomes of Gynecological Oncology Patients at Assiut University: A Retrospective Study (2022-2025)
Brief Title: Survival Outcomes of Gynecologic Oncology Patients at Assiut University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Farouk, Resident at Obstetric and Gynecology Department, Assiut University
Other Study IDs: Gynecological Oncology Outcome
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Gynaecological Oncology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This retrospective cohort study investigates survival outcomes of gynecological oncology patients treated at Assiut University Hospital between 2022 and 2025, comparing them to international benchmarks and assessing factors affecting survival.

DETAILED DESCRIPTION:
The study aims to evaluate overall survival (OS) and progression-free survival (PFS) of patients diagnosed with gynecological cancers (including ovarian, cervical, endometrial, vulvar, and vaginal cancers) and treated at Assiut University Hospital from January 1, 2022, to December 31, 2025. Using retrospective medical records and pathology reports, the study will analyze demographic, clinical, and treatment-related variables to identify factors influencing survival outcomes. Assiut University is a tertiary care center in a low-resource setting; thus, the study will also assess adherence to international oncology guidelines (e.g., ESMO, ASCO) and compare local survival rates with international standards. Statistical methods include Kaplan-Meier survival analysis and Cox proportional hazards modeling.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with gynecological cancers (ovarian, cervical, endometrial, vulvar, vaginal)

Patients treated at Assiut University Gynecological Oncology Department between January 1, 2022, and December 31, 2025

All age groups included

Exclusion Criteria:

- Patients with non-gynecological malignancies or metastatic cancers originating outside the gynecological tract

Patients with incomplete medical records (e.g., missing pathology reports or treatment details)

Patients with significant comorbidities independently affecting survival (e.g., advanced heart failure, severe liver or renal disease, terminal illnesses unrelated to cancer)

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All female patients diagnosed with gynecological cancers (including ovarian, cervical, endometrial, vulvar, and vaginal cancer) and treated at Assiut University Gynecological Oncology Department between January 1, 2022, and December 31, 2025, will be included. Patients of all ages and backgrounds are eligible. Exclusion criteria are non-gynecological cancers, metastatic cancers originating outside the gynecologic tract, incomplete medical records, or significant comorbidities that independently affect survival (e.g., advanced heart failure, severe liver or renal disease, or unrelated terminal illnesses).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4 years
  Overall survival (OS) is defined as the duration of time from the date of cancer diagnosis or initiation of treatment until death from any cause. Patients will be censored at the date of last follow-up if alive at study end. This outcome will provide a direct estimate of survival rates among gynecological oncology patients treated at Assiut University Hospital.